CLINICAL TRIAL: NCT02502201
Title: Effect of the Environment on Six-minute Walk Test Performance in Individuals With Alpha-1 Antitrypsin Deficiency-Related Chronic Obstructive Pulmonary Disease
Brief Title: Environment Effect on Six-Minute Walk Test Performance
Acronym: 6MWTAATD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty finding participants who fit all criteria
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201500220
Record Dates: First submitted 2015-06-09; First posted 2015-07-20 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Alpha-1 Antitrypsin Deficiency
Keywords: six-minute walk
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- six-minute walk study indoors first (Active Comparator): Participants randomized to indoor six-minute walk test first
  Interventions: Other: six-minute walk study indoors
- six-minute walk study outdoors first (Experimental): Participants randomized to outdoor six-minute walk test first
  Interventions: Other: six-minute walk study outdoors
- six-minute walk study indoors second (Active Comparator): Participants randomized to indoor six-minute walk test second
  Interventions: Other: six-minute walk study indoors
- six-minute walk study outdoors second (Experimental): Participants randomized to outdoor six-minute walk test second
  Interventions: Other: six-minute walk study outdoors

INTERVENTIONS:
Other: six-minute walk study indoors — Performance of a six-minute walk test according to American Thoracic Society standard.
  Arms: six-minute walk study indoors first; six-minute walk study indoors second
Other: six-minute walk study outdoors — Performance of a six-minute walk test.
  Arms: six-minute walk study outdoors first; six-minute walk study outdoors second

SUMMARY:
The purpose of this research study is to determine the effect of the environment on six-minute walk test performance in individuals with chronic obstructive pulmonary disease due to alpha-1 antitrypsin deficiency. The aim of the study is to determine the environmental impact on physical performance in this population to determine if any factors influence quality of life. This study was developed to evaluate the efficacy of the using the indoor six-minute walk test to determine eligibility for ambulatory oxygen therapy.

DETAILED DESCRIPTION:
Participants will be asked to come to the Clinical Research Center (CRC) for a visit lasting about one hour. Participants will be asked to review and sign an informed consent document to participate in this trial. If participants agree to participate and sign the consent, the following procedures will be done. If they have not had pulmonary function testing performed in the past 18 months, standard spirometry testing will be performed. Participants will perform two six-minute walk tests, one indoors and one outdoors. First, they will be randomly assigned to perform either the indoor or outdoor testing first. Then participants will have their vital signs taken, perform the first six-minute walk study and immediately after have their vital signs taken again. Participants will have a rest period between the two six-minute walk tests of at least 30 minutes. Participants will then perform the second six-minute walk test with the same above procedures for the first test.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Have a diagnosis of congenital Alpha-1 Antitrypsin Deficiency with an allelic combination of ZZ.
3. Have a Forced Expiratory Volume in 1 second (FEV1)< 50% of predicted and FEV1/forced vital capacity (FVC) < 70% (Global Initiative for Chronic Obstructive Lung Disease [GOLD] stage II, III, or IV).
4. Not currently prescribed Oxygen replacement at a rate of greater than 2 liters.
5. Willing and able to perform two six-minute walk tests.
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Subject has had a moderate or severe pulmonary exacerbation during the 4 weeks before the study visit.
2. History of lung transplant.
3. Severe concomitant disease (e.g., congestive heart failure, clinically significant pulmonary fibrosis, malignant disease [with the exception of skin cancers other than melanoma], history of acute hypersensitivity pneumonitis reaction, or current chronic hypersensitivity pneumonitis).
4. Unwilling or unable to perform six-minute walk testing.
5. Mentally challenged adult subjects who cannot give independent informed consent.
6. In the opinion of the investigator the subject may have compliance problems with the protocol and the procedures of the protocol.
7. American Thoracic Society listed absolute contraindications to six-minute walk test: unstable angina or myocardial infarction during previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change in the meters walked during the six-minute walk test between the two groups. | baseline

SECONDARY OUTCOMES:
Change in Borg Scale for shortness of breath between the two groups | baseline
  The Borg Scale a numerical scale for assessing shortness of breath, from 0 representing no shortness of breath to 10 as maximal shortness of breath.
Change in Borg Scale for fatigue between the two groups | baseline
  The Borg Scale a numerical scale for assessing shortness of breath, from 0 representing no shortness of breath to 10 as maximal shortness of breath.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brantly, MD, Principal Investigator — University of Florida
Locations (1):
- Uf Ctsi Crc, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No